CLINICAL TRIAL: NCT07039747
Title: Effectiveness of a Dietary Supplement in Irritable Bowel Syndrome
Acronym: ACALMI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Laboratoire Dielen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/0178/HP
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: glutamine
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment with DIELEN® Protect (Experimental): experimental group: treatment with DIELEN® Protect for 8 weeks at a dose of 5 grams, 3x a day
  Interventions: Drug: treatment with DIELEN® Protect
- control group (Placebo Comparator): Control group: treatment with placebo (pea protein) for 8 weeks at a dose of 5 grams, 3x a day
  Interventions: Drug: treatment with placebo of DIELEN® Protect

INTERVENTIONS:
Drug: treatment with DIELEN® Protect — treatment with DIELEN® Protect for 8 weeks at a dose of 5 grams, 3x a day
  Arms: treatment with DIELEN® Protect
Drug: treatment with placebo of DIELEN® Protect — treatment with placebo of DIELEN® Protect for 8 weeks at a dose of 5 grams, 3x a day
  Arms: control group

SUMMARY:
Irritable bowel syndrome (IBS) affects around 5% of the general population and remains a daily problem in clinicians' practices, with inconsistent efficacy of treatments despite patients' high expectations. Intestinal hyperpermeability and visceral hypersensitivity are the two major components of IBS, and both can disrupt gastrointestinal function and ultimately impair patients' quality of life.

Glutamine is a non-essential amino acid that regulates numerous metabolic pathways and plays a key role in the intestine as it is the preferred substrate for enterocytes and immune cells. A decrease in intestinal glutamine synthetase has been found in IBS, suggesting its involvement in the intestinal permeability and visceral hypersensitivity observed in patients. Ex vivo, glutamine is capable of restoring the expression of tight junction proteins in IBS-D patients. Furthermore, glutamine supplementation is capable of reducing abdominal pain and restoring intestinal permeability disorders in a sub-group of patients with intestinal permeability disorders (post-infectious IBS-D).

The marine peptides Gabolysat® produced by the Dielen Laboratory have demonstrated their efficacy on intestinal permeability and inflammation in a preclinical model of IBS (Langlois et al. 2023), similar to glutamine supplementation in these animals. The Dielen® Protect product formulated on the basis of the results of this study combines glutamine and Gabolysat® to provide a comfort solution for IBS patients.

Our working hypothesis is that patients suffering from moderate or severe IBS could benefit from oral supplementation with DIELEN Protect to improve the symptoms associated with IBS.

100 patients with IBS (according to Rome IV criteria) will be included in our study.

All patients will test the treatment for 8 weeks (dielen protect or placebo). The efficacy will be compared between the 2 groups before and after the treatments using validated questionnaires. Therefore, all participants will fill questionnaire before and after 8 weeks of treatments : IBS severity (IBS-SSS), quality of life (GIQLI), Anxiety and depression (HAD), GI symptom related anxiety (VSI), stool frequency and consistancy (BSF scale). Microbiota, metabolomic and short chain fatty acid will be analysed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Irritable bowel syndrome according to Rome IV criteria
* Aged between 18 and 75 years
* IBS-SSS > 175 at inclusion
* For women of childbearing age, use of effective contraception (progestins or oestroprogestins or intrauterine device or tubal ligation) for 1 month unless postmenopausal (amenorrhoea of at least 12 months or biologically confirmed diagnosis) or woman who has had a hysterectomy or salpingectomy.
* Irritable bowel syndrome treatments that have been stable for more than one month
* Membership of a social security scheme
* Patient has read and understood the information letter and signed the consent form

Exclusion Criteria:

* Taking probiotics, food supplements containing glutamine, anti-inflammatory drugs or antibiotics in the month preceding the study.
* Allergy to fish and glutamine
* Known renal insufficiency (Glomerular Filtration Rate (GFR)<30mL/min/1.73m2), known hepatic insufficiency (Prothrombin Time (PT)<70%) or known cardiac disease.
* History of organic digestive disease (coeliac disease, inflammatory bowel disease, abdominal surgery other than appendectomy or cholecystectomy)
* Pregnant women, women in labour or breastfeeding mothers
* Person deprived of liberty by an administrative or judicial decision or person placed under court protection / sub-guardianship or guardianship
* Patient taking part in another trial / having taken part in another trial within a 4-week period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Symptomatic efficacy of DIELEN® Protect supplementation | from enrollment up to 8 weeks
  change in IBS severity score (IBS-SSS) measured before and after 8 weeks of DIELEN® Protect or placebo supplementation in patients The IBS-SSS is a questionnaire used to assess the severity of irritable bowel syndrome.

SECONDARY OUTCOMES:
impact of DIELEN® Protect on the composition of the intestinal microbiota | from enrollment up to 8 weeks
  variation in the composition of faecal microbiota measured before and after supplementation with DIELEN® Protect or placebo for 8 weeks.
Impact of DIELEN® Protect on quality of life | from enrollment up to 8 weeks
  change in GIQLI score measured before and after 8 weeks' supplementation with DIELEN® Protect or placebo GILQLI : self-administered questionnaire completed by the patient, comprising 36 questions relating to digestive symptoms, their social and emotional impact, and general condition over the last few days. The answer to each question is scored from 0 (permanent symptoms) to 4 (no symptoms). The individual score is calculated by adding up all the points obtained for all the items. The overall score varies from 0 (worst possible quality of life) to 144 (best possible quality of life).
impact of DIELEN® Protect on gastrointestinal related anxiety | from enrollment up yto 8 weeks
  change in VSI score measured before and after DIELEN® Protect or placebo supplementation for 8 weeks
  VSI : 'gastrointestinal related anxiety' scale. This scale is based on 15 questions, all with answers ranging from 0 to 5. At the end of the questionnaire, a score out of 75 is obtained. Scores close to 0 indicate no gastrointestinal anxiety, while scores close to 75 indicate severe gastrointestinal anxiety.
impact of DIELEN® Protect on anxiety and/or depression | from enrollment up to 8 weeks
  variation in HAD score measured before and after 8 weeks' supplementation with DIELEN® Protect or placebo
  The HAD scale detects the presence of anxiety or depression. Each symptom is scored on 21 points. A score below 8 eliminates anxiety or depression, a score between 8 and 10 defines a doubtful state of anxiety or depression, and a score above 10 a definite state of anxiety or depression.
impact of DIELEN® Protect on stool frequency | from enrollment up to 8 weeks
  variation in the mean number of stools per day before and after 8 weeks' supplementation with DIELEN® Protect or placebo (stool calendar)
impact of DIELEN® Protect on stool consistency | from enrollment up to 8 weeks
  variation in the Bristol stool form before and after 8 weeks' supplementation with DIELEN® Protect or placebo
  the Bristol stool form (Score de Bristol) class stools in 7 types from type 1 = constipation to type 7 = diarrhoea
treatment compliance | from enrollment up tu 8 weeks
  Compliance will be assessed by measuring the number of sachets of DIELEN® Protect or placebo not taken after 8 weeks of treatment. The patient will be considered non-compliant if the uptake of DIELEN® Protect or placebo over the 8 weeks is < 70%.
treatment tolerance | from enrollment up to 8 weeks
  Tolerance will be assessed by the number and severity of adverse reactions at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chloé MELCHIOR, PUPH, Principal Investigator — University Hospital, Rouen
Locations (1):
- CHU de Rouen, Rouen, France, France

IPD SHARING:
Plan to Share IPD: Undecided